CLINICAL TRIAL: NCT03399604
Title: A Phase 3 Open-label, Multicenter Study to Evaluate the Long-term Safety and Tolerability of Inhaled LIQ861(Treprostinil) in Pulmonary Arterial Hypertension (WHO Group 1) Patients
Brief Title: Investigation of the Safety and Pharmacology of Dry Powder Inhalation of Treprostinil
Acronym: INSPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Liquidia Technologies, Inc. (Industry)
Collaborators: Nuventra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTI-301
Record Dates: First submitted 2018-01-03; First posted 2018-01-16 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Primary Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension; Idiopathic Pulmonary Arterial Hypertension; Heritable Pulmonary Arterial Hypertension; Drug Induced Pulmonary Arterial Hypertension; Toxin Induced Pulmonary Arterial Hypertension; Connective tissue disease
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Pulmonary Arterial Hypertension; Connective Tissue Diseases

STUDY DESIGN:
Intervention Model Description: The study will evaluate the long term safety and tolerability of LIQ861 in PAH patients transitioning from stable doses of inhaled treprostinil therapy, or who are taking no more than 2 approved, non-prostacylcin, oral PAH therapies.
  Patients transitioning from inhaled treprostinil will be initiated at a comparable dose of LIQ861, and then titrate in 25ug incremental doses to tolerance and symptom relief. Patients adding LIQ861 to current oral therapies will start at a 25ug dose, and increase in 25ug increments on a weekly basis to tolerance and symptom relief.
  A subset of the patients transitioning from inhaled treprostinil will be enrolled in a one-directional crossover to compare the bioavailability and pharmacokinetics of treprostinil as they transition to LIQ861. Serial PK sample collections will be taken on back to back days for transitioning and LIQ861 treprostinil formulations. These patients will then continue to be followed as all other patients enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LIQ861 Inhaled Treprostinil (Experimental): LIQ861 inhaled treprostinil at capsule strengths of 25 μg, 50 μg, 75 μg and 100 μg.
  LIQ861 will be administered using the RS00 Model 8 dry powder inhalation (DPI) device (Plastiape S.p.A.; Osnago, Italy) at dose levels of 25 μg to 150 μg treprostinil QID in individual patients.
  Interventions: Drug: LIQ861 Inhaled Treprostinil

INTERVENTIONS:
Drug: LIQ861 Inhaled Treprostinil — LIQ861 bulk powder is generated from a treprostinil/excipient matrix from which particles of precise size and shape are created and filled into a hydroxypropyl methylcellulose (HPMC) capsule (size 3). LIQ861 capsules are provided in capsule strengths of 25 μg, 50 μg, 75 μg and 100 μg treprostinil.
  Other Names: inhaled treprostinil; inhaled prostacyclin

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of LIQ861, a dry powder formulation of treprostinil, in patients with Pulmonary Arterial Hypertension (PAH).

DETAILED DESCRIPTION:
One of the greatest impediments to patient treatment satisfaction with current inhaled treprostinil therapy is inconvenience. Currently, PAH patients using inhaled treprostinil may require more than 36 breaths per day using a nebulizer requiring daily set up and cleaning. The use of a discrete, hand-held dry powder inhaler to deliver treprostinil to the lungs could represent a major improvement in convenience and patient satisfaction, thereby improving the quality of life for PAH patients. Liquidia is pursuing approval of LIQ861, an inhalation dry powder formulation of treprostinil that is produced using Liquidia's PRINT® Technology (Particle Replication in Nonwetting Templates), as an alternative to current inhaled treprostinil therapy for the treatment of patients with PAH (WHO Group 1).

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent by patient prior to study enrollment
* 18 years of age or older
* If female of childbearing potential, a negative pregnancy test at the Baseline Visit and agrees to practice adequate birth control throughout the duration of the study. If the patient is postmenopausal or has documented surgical sterilization, a pregnancy test and birth control is not necessary.
* The patient has been diagnosed with PAH belonging to the following subgroups of the updated Nice Clinical Classification Group 1 (Simonneau, Gatzoulis et al. 2013), which include:

  1. Idiopathic PAH (1.1), or
  2. Heritable PAH (1.2), or
  3. Drug and toxin induced PAH (1.3), or
  4. PAH associated with connective tissue disease (1.4.1), HIV infection (1.4.2), or congenital heart disease (1.4.4) with simple systemic-to-pulmonary shunt at least 1 year after surgical repair
* The patient has been diagnosed with PAH and is NYHA Functional Class II - IV at Screening.

  1. has documented stable doses of approved inhaled therapy for at least 3 months prior to screening and is willing and able to transition from their prescribed dose of inhaled therapy to study drug, or
  2. has documented stable doses of no more than two approved oral therapies for at least 3 months prior to screening and is willing and able to add LIQ861 to their treatment regimen.
* The patient can complete a baseline six-minute walk distance (6MWD) ≥ 150 m.
* The patient has had evidence of FEV1 ≥ 60% and FEV1/FVC ratio ≥ 60% during the 6-month period prior to enrollment.

Exclusion Criteria:

* The patient's clinical condition is such that, in the opinion of the Investigator, they are not expected to remain clinically stable for the duration of the study.
* Patients with PH in the Updated Nice Classification Groups 2-5, or PAH Group 1 subgroups not covered by the inclusion criteria (e.g., associated with portal hypertension [1.4.3] or with schistosomiasis [1.4.5]).
* The patient is currently taking oral prostacyclin analogues or agonists, including treprostinil and selexipag.
* The patient has had any PAH medication (except for anticoagulants) discontinued within 14 days of Baseline.
* The patient has had a new type of chronic therapy (including but not limited to oxygen, a different class of vasodilator, diuretic, digoxin, and digitalis) for pulmonary hypertension added within 30 days of Baseline.
* The patient has uncontrolled systemic hypertension as evidenced by persistent systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg.
* The patient has a history of hemodynamically significant left-sided heart disease including, but not limited to: aortic or mitral valve disease, pericardial constriction, restrictive or congestive cardiomyopathy, or coronary artery disease (CAD).
* The patient has had an atrial septostomy.
* The patient has any serious or life-threatening disease other than conditions associated with PAH (e.g. malignancy requiring aggressive chemotherapy, end stage renal disease, etc.).
* The patient is taking any excluded medications listed in the Investigator's Brochure, namely inhibitors and inducers of CYP2C8
* The patient has a hypersensitivity or allergy to any of the ingredients of LIQ861 or other clinically relevant allergies (clinical relevance per Investigator judgment).
* The patient has had a pulmonary infarction (defined as infarction in more than one lung segment documented by V/Q scan or pulmonary angiography) within two weeks of Screening.
* The patient has had a stroke or transient ischemic attack (TIA) within six months of Screening.
* The patient has evidence of an active uncontrolled sepsis or systemic infection during Screening.
* The patient is pregnant or lactating.
* The patient has any musculoskeletal disease or any other disease that would limit ambulation.
* The patient has participated in an investigational product or device study within the 30 days prior to Screening.
* The patient has current evidence of drug abuse in the opinion of the Investigator.
* The patient has severe hepatic impairment as evidenced by any history of ascites AND encephalopathy.
* The patient has severe renal impairment (eGFR < 35).
* The patient is taking inhaled treprostinil doses of greater than 90 μg (more than 15 breaths).

Additional Exclusion Criteria for PK Sub-Study:

* The patient meets any of Primary Exclusion Criteria #1 - 19.
* The patient has moderate or severe renal impairment (eGFR < 60).
* The patient is taking inhaled treprostinil doses of greater than 72 μg (more than 12 breaths).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Hill, MD, Principal Investigator — Tufts Medical Center
Locations (38):
- United States (38):
  - Banner University Medical Center, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Los Angeles Biomedical Research Center, Torrance, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth, Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Wellstar Research Institute, Marietta, Georgia
  - Northwestern Medicine, Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kentuckiana Pulmonary Research Center, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - NYU Winthrop University Hospital, Mineola, New York
  - NYU Langone Health, New York, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals of Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - the Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science Center, Portland, Oregon
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Alleghany General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Lung Center, Houston, Texas
  - University of Texas - Health Science Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - INOVA Fairfax Medical Campus, Falls Church, Virginia
  - The Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roscigno R, Vaughn T, Anderson S, Wargin W, Hunt T, Hill NS. Pharmacokinetics and tolerability of LIQ861, a novel dry-powder formulation of treprostinil. Pulm Circ. 2020 Nov 19;10(4):2045894020971509. doi: 10.1177/2045894020971509. eCollection 2020 Oct-Dec. PMID 33282202

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 146 subjects screened for the study, 121 (55 Transition Group, 66 Add On Group) were enrolled.
Groups:
- LIQ861 Inhaled Treprostinil: LIQ861 inhaled treprostinil at capsule strengths of 25 μg, 50 μg, 75 μg and 100 μg.
  LIQ861 will be administered using the RS00 Model 8 dry powder inhalation (DPI) device (Plastiape S.p.A.; Osnago, Italy) at dose levels of 25 μg to 150 μg treprostinil QID in individual patients.
  LIQ861 Inhaled Treprostinil: LIQ861 bulk powder is generated from a treprostinil/excipient matrix from which particles of precise size and shape are created and filled into a hydroxypropyl methylcellulose (HPMC) capsule (size 3). LIQ861 capsules are provided in capsule strengths of 25 μg, 50 μg, 75 μg and 100 μg treprostinil.
Period: Overall Study
Arm/Group | LIQ861 Inhaled Treprostinil
Started | 121
Completed | 92
Not Completed | 29

BASELINE CHARACTERISTICS:
Population: All enrolled subjects were included in the Safety Population. The Efficacy Population included all but 1 subject (who had no post-Baseline efficacy assessments performed and was lost to follow-up. The mITT Population, which included all subjects identified as WHO Group 1 based upon adjudication by a panel of PAH experts, comprised 106 subjects. The PK Population included 18 subjects in the Transition Group.
Arm/Group | LIQ861 Inhaled Treprostinil
Number analyzed (Participants) | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 95
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 15
  White | 96
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 121

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events and Serious Adverse Events
Description: There were two treatment arms analyzed for events in the study. All subjects that participated in the PK study were part of the transition group and not analyzed separately for adverse events.
  Treatment-Emergent Adverse Events and Serious Adverse Events will be grouped by MedDRA System Organ Class, dose level, time on drug, and relationship to dose titration
Time Frame: Baseline, Week 2, Month 1, Month 2 Visits, with bimonthly follow up for up to 16 months.
Population: The Safety Population included all subjects who received at least 1 inhalation of LIQ861.
Measure: Count of Participants; unit: Participants
Arm/Group | LIQ861 Inhaled Treprostinil
Number analyzed (Participants) | 121
Participants | 121

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Groups:
- LIQ861 Add-On: LIQ861 inhaled treprostinil at capsule strengths of 25 μg, 50 μg, 75 μg and 100 μg.
  LIQ861 will be administered using the RS00 Model 8 dry powder inhalation (DPI) device (Plastiape S.p.A.; Osnago, Italy) at dose levels of 25 μg to 150 μg treprostinil QID in individual patients.
  LIQ861 Inhaled Treprostinil: LIQ861 bulk powder is generated from a treprostinil/excipient matrix from which particles of precise size and shape are created and filled into a hydroxypropyl methylcellulose (HPMC) capsule (size 3). LIQ861 capsules are provided in capsule strengths of 25 μg, 50 μg, 75 μg and 100 μg treprostinil.
- Tyvaso Transition: LIQ861 inhaled treprostinil at capsule strengths of 25 μg, 50 μg, 75 μg and 100 μg.
  LIQ861 will be administered using the RS00 Model 8 dry powder inhalation (DPI) device (Plastiape S.p.A.; Osnago, Italy) at dose levels of 25 μg to 150 μg treprostinil QID in individual patients.
  LIQ861 Inhaled Treprostinil: LIQ861 bulk powder is generated from a treprostinil/excipient matrix from which particles of precise size and shape are created and filled into a hydroxypropyl methylcellulose (HPMC) capsule (size 3). LIQ861 capsules are provided in capsule strengths of 25 μg, 50 μg, 75 μg and 100 μg
Arm/Group | LIQ861 Add-On | Tyvaso Transition
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/121
Serious Adverse Events (participants affected / at risk) | 15/121 | 6/121
Other Adverse Events (participants affected / at risk) | 66/121 | 55/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LIQ861 Add-On (N=121) | Tyvaso Transition (N=121)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Acute on Chronic Hypoxic Respiratory Failure
Cardiac Failure (Cardiac disorders) | 1 (1) | 1 (1) — Worsening Volume Overload
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Worsening of PAH
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Struma Ovarii
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Possible Hypersensitivity Pneumonitis
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Atrial Fibrillation Exacerbation
Pyrexia (General disorders) | 1 (1) | 0 (0) — Fever
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Worsening Hypoxia
Diaphragmatic Paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Left Hemidiaphragmatic Paresis
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) — Possible Pneumonia
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Worsening of Shortness of Breath
Syncope (Nervous system disorders) | 2 (2) | 0 (0) — Syncope
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0) — Hypertensive Urgency
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) — Viral Illness
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — Sepsis
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) — Acute Kidney Injury
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — Possible Seizure Activity
Parainfluenzae Virus Infection (Infections and infestations) | 1 (1) | 0 (0) — Parainfluenzae
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Acute on Chronic Hypoxic Respiratory Failure
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — Non ST Elevation Myocardial Infarction
Open Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Compound Fracture of Lower Leg
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) — Worsening Lower Extremity Edema
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0) — Worsening Left Internal Carotid Stenosis
Fluid Overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Fluid Overload
Overgrowth Bacterial (Infections and infestations) | 0 (0) | 1 (1) — Exacerbation of Chronic Bacterial Overgrowth
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Pulmonary Embolism
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — GI Bleed
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LIQ861 Add-On (N=121) | Tyvaso Transition (N=121)
Cough (Respiratory, thoracic and mediastinal disorders) | 41 (41) | 23 (23) — Cough
Dysponea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 13 (13)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 23 (23) | 18 (18)
Dizziness (Nervous system disorders) | 13 (13) | 10 (10)
Upper Respiratory Tract Infection (Infections and infestations) | 18 (18) | 10 (10)
Nasopharyngitis (Infections and infestations) | 6 (6) | 6 (6)
Urinary Tract Infection (Infections and infestations) | 6 (6) | 2 (2)
Chest Discomfort (General disorders) | 7 (7) | 11 (11)
Fatigue (General disorders) | 10 (10) | 4 (4)
Pyrexia (General disorders) | 7 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Flushing (Vascular disorders) | 7 (7) | 3 (3)
Diahrrea (Gastrointestinal disorders) | 15 (15) | 7 (7) — Diarrhea
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6) — Nausea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03399604/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT03399604/SAP_001.pdf